CLINICAL TRIAL: NCT01940042
Title: the Effect of Simple Clinical Maneuver on Shoulder and Abdominal Pain a Laparascopic Gynecological Surgery:a Prospective Randomised Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bakirkoy Maternity and Children Diseases Hospital (Other Government)
Responsible Party: Principal Investigator, Osman Aşıcıoğlu, Medical Doctor, Istanbul Bakirkoy Maternity and Children Diseases Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: aşıcıoğlu07
Record Dates: First submitted 2013-09-07; First posted 2013-09-11 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Effect of CO2 Was Removed by Means Trandelenburg Position at Laparascopic Surgery

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- maneuver group (Experimental): In the intervention group, CO2 was removed by means of Trendelenburg position (30 degrees) and a pulmonary recruitment maneuver consisting of five manual inflations of the lung.
  Interventions: Behavioral: CO2 was removed by means of trandelenburg positions
- clasical group (No Intervention): no additional action will be taken after the operation

INTERVENTIONS:
Behavioral: CO2 was removed by means of trandelenburg positions
  Arms: maneuver group

SUMMARY:
The investigators think that a simple maneuver at laparascopic surgery to reduce the postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

1. females aged 15-65 years,
2. American Society of Anesthesiologists (ASA) physical status classification I-III
3. no previous laparotomy(major abdominal surgery).
4. need a laparascopic surgery

Exclusion Criteria:

1. required hospitalization after the laparoscopic surgery,
2. the procedure required conversion to laparotomy
3. if a 48-hour follow-up was not feasible

Ages: 15 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
postoperative 12. hour VAS pain score | 12 hour

SECONDARY OUTCOMES:
postoperative analgesic requırements | 48 hours

OTHER OUTCOMES:
postoperative shoulder pain score | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: isa aykut özdemir, m.d., Principal Investigator — tepecik education and research hospital
Locations (1):
- Tepecik Education and Research Hospital, Izmir, Turkey (Türkiye)

REFERENCES:
- [Result] Esin S, Culha ZK, Kara OF, Yildirim H. A simple clinical maneuver to reduce laparoscopy-induced shoulder pain: a randomized controlled trial. Obstet Gynecol. 2008 Aug;112(2 Pt 1):380; author reply 380. doi: 10.1097/AOG.0b013e318182cb6e. No abstract available. PMID 18669740
- [Derived] Gungorduk K, Asicioglu O, Ozdemir IA. Effect of the pulmonary recruitment maneuver on pain after laparoscopic gynecological oncologic surgery: a prospective randomized trial. J Gynecol Oncol. 2018 Nov;29(6):e92. doi: 10.3802/jgo.2018.29.e92. PMID 30207100